

## Effect of Bilateral Distalization of Upper First Molars in a Group of Patients after extraction of Maxillary Second Molars Using Infra Zygomatic Mini Implants Prospective clinical trial

### Consent Form

Faculty of Dentistry, Future University in Egypt

## Submitted by

Name: Hosam Abdullah Mohamed Zaza

B.D.S. Future University, 2017 (2020)

| | Document is approved for use by the ics Committee of FUE/FODM |
|------------|---------------------------------------------------------------|
| Date From: | |
| To: | |



# RESEARCH ETHICS COMMITTEE Faculty of Oral and Dental Medicine (REC-FODM)

CONSENT FORM (#3)

#### Title of Research:

Effect of Bilateral Distalization of Upper First Molars in a Group of Patients after extraction of Maxillary Second Molars Using Infra Zygomatic Mini Implants Prospective clinical trial

# **Part I – Research Participant Information Sheet:**

- **A.** Purpose of the Research is to evaluate the dentoalveolar effect of the infrazygomatic mini implant supported destalizer when used for bilateral distalization of the maxillary molars.
- **B.** Description of the Research: this trial will involve distalization of maxillary first molars using infra-zygomatic mini implant supported appliance to correct class II malocclusion.
- C. Potential Risks and Discomforts: pain associated with tooth movement, inflammation of mucosal tissues
- D. Potential Benefits: orthodontic treatment is done for the patient as indicated, improving patients' esthetics, function and psychology including protrusion.

| This Consent Document is approved for use by the Research Ethics Committee of FUE/FODM | |
|---|---|
| REC # : | |
| Date From: | _ |
| To: | |



- E. Cost: To participate in the research you will bear no additional costs or extra loss.
- F. Compensation / Treatment:

In the event of injury resulting from participation in this research study, Researcher will make a treatment to you, its facilities and professional attention. Financial compensation from FUE/FODM is not available.

#### **G.** Voluntary Participation:

Participation in this study is voluntary. You will suffer no penalty nor loss of any benefits to which you are otherwise entitled should you decide not to participate. Withdrawal from this research study will not affect your ability to receive alternative methods of Dental care available at FUE/FODM. Significant new findings developed during the course of the research study which might be reasonably expected to affect your willingness to continue to participate in the research study will be provided to you.

#### H. Confidentiality:

Your identity and medical record, as a participant in this research study, will remain confidential with respect to any publications that may result from this study. Furthermore, your Dental/medical record may be reviewed by the Research Advisory Council or the agency sponsoring this research in accordance with applicable laws and regulations.

| I. | Contact Person(s): | |
|----|----------------------------------------------------|-----|
| | signed copy of the consent form will be given you. | vei |

| Fhis Consent Document is approved for use by the Research Ethics Committee of FUE/FODM REC #: |
|---|
| Date From: |
| To: |



# PART II - Authorization for performance of certain procedures:

- 1. I/surrogate authorize Dr. Hosam Abdullah Zaza and her associates to administer the following drugs, use the following devices or perform the following procedures during my treatment (or the treatment of the person named above for whom I am responsible)
- 2. I acknowledge that I have read, or had explained to me in a language I understand, the attached Research Participant Information sheet and that Dr. Hosam Abdullah Zaza has explained to me the nature of the procedures described in the Research Participant Information Sheet as well as any benefits to be expected, possible alternative methods of treatment, the attendant discomforts and risks reasonably to be expected and the possibility that complications from both known and unknown causes may arise as a result thereof. I was given ample opportunity to comprehensively inquire about this study and procedures and all my questions were answered to my satisfaction.
- 3. I understand that I am not entitled for reimbursement for expenses incurred as a result of my participation in this study

| This Consent Document is approved for use by the Research Ethics Committee of FUE/FODM REC #: | |
|---|---|
| Date From: | _ |
| To: | |



- 4. I voluntarily accept the risks associated with the above-mentioned procedures with the knowledge and understanding that the extent to which they may be effective in my treatment (or the treatment of the patient named above, as the case may be) has not been established, that there may be side effects and complications from both known and unknown causes and that these procedures may not result in cure or improvement.
- 5. I understand that I am free to withdraw this consent and discontinue treatment with the above procedures at any time. The consequences and risks, if any, which might be involved in the event I later decide to discontinue such treatment, have been explained to me adequately. I understand that such withdrawal will not affect my ability to receive any dental/medical care made necessary by the performance of such studies or to which I might be otherwise entitled.

6. I confirm that I have read, or had read to me,

the foregoing authorization and that all blanks or statements requiring completion were properly completed before I signed.

Patient
Name:
File #:
Patient/Surrogate:

Signature

Date

Relationship:

| | Document is approved for use by the ics Committee of FUE/FODM |
|------------|---------------------------------------------------------------|
| Date From: | |
| To: | |



**Research Ethics Committees** 

Faculty of Oral and Dental Medicine
7. I confirm that I have accurately translated and/or read the information to the subject or his/her surrogate.

| Name: | |
|---|---|
| Signature: | |
| FUE ID #:<br>Date: | |
| 8. I have fully explained to the above p relative/ guardian the nature and purpo foregoing procedures, possible alternative methods of treatment which might be advantageous, the reasonable benefits to expected, the attendant discomforts and involved, the possibility that complication arise as a result thereof and the consequent and risks, if any, which might be involved event the patient/ relative/ guardian here decides to discontinue such treatment. It is my understanding that the above parelative/ guardian understand the nature purposes, benefits, and risks of participathis research before signing of this infor consent. I have also offered to answer a questions the above patient/ relative/ guardian that the above patient relative guardian that the above patient relative guardian that the above patient relative guardian that the above patient relative guardian that also offered to answer a questions the above patient answered all squestions. | se of the ve be risks ons may ences ed in the eafter atient/ e, ation in med ny ardian ures and |
| (Signature of Principal Investigator/ Del | legate): |
| Print Name: Hosam Abdullah Mohamed | d Zaza |
| Title: Master Student at FUE. | |

This Consent Document is approved for use by the Research Ethics Committee of FUE/FODM REC #:\_ Date From: To:\_